CLINICAL TRIAL: NCT06326645
Title: Open-Label Pilot Study With Crofelemer in Patients With Short Bowel Syndrome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lindsey Russell, MD (Other)
Collaborators: Napo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lindsey Russell, MD, Staff Gastroenterologist, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-891
Record Dates: First submitted 2023-11-25; First posted 2024-03-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Short Bowel Syndrome
Keywords: SBS
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Small exploratory study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Crofelemer Group (Experimental)
  Interventions: Drug: Crofelemer Oral Product

INTERVENTIONS:
Drug: Crofelemer Oral Product — Crofelemer powder for solution (50g and 100g) or Crofelemer Powder for Oral Solution (100 mg/mL or 30 mg/mL vials for reconstitution and oral dosing)

SUMMARY:
The objectives of this study are to evaluate the efficacy and safety of crofelemer treatment in adults affected by Short Bowel Syndrome (SBS) with an ileostomy on parenteral support (PS) in reducing output or PS needs. Crofelemer will be provided as a powder three times daily for 12 weeks and a 4 week follow up. .

DETAILED DESCRIPTION:
Short bowel syndrome (SBS) is defined as less than 200 cm in adults of remaining small bowel (i.e. excluding colon) in continuity leading to the need for nutritional and fluid supplements due to impaired absorption of nutrients, electrolytes and fluids.

Most patients with SBS experience debilitating diarrhea that severely hinders their health outcomes and quality of life. SBS-associated diarrhea may have several etiologies including excessive secretion and/or impaired absorption of fluid and electrolytes across the intestinal epithelium. Diarrhea can lead to dehydration, electrolyte imbalance, protein-calorie malnutrition, and loss of critical vitamins and minerals. Consequently, diarrhea in SBS can be severe and life-threatening without proper treatment.

The aggressive use of anti-diarrheal medications in SBS are often clinically required to help manage symptoms. Anti- Secretory agents, including proton pump inhibitors, histamin-2 receptor agonists and somatostatin analogue (Octreotide) as well as various anti-motility agents, including loperamide, Diphenoxylate/atropine, and opioids (Codeine, Tincture of Opium), are often used in higher doses and various formulations with varying effects in patients to help control the diarrhea. Overall, the management of diarrhea is challenging requiring multidisciplinary teams and improved therapies are needed.

Parenteral Nutrition (PN) is a life-saving therapy for patients unable to meet nutritional needs by mouth and a recent study noted that SBS is the most common indication for home PN in the US. However, long-term PN is associated with experience serious metabolic complications, including hepatic and biliary disorders manifested by steatosis, fibrosis and cholestasis. Other complications include central line infections and decrease in quality of life. This has garnered orphan drug designation for intestinotrophic hormones like the glucagon-like peptide-2 (GLP-2) analogue, teduglutide (Gattex), which increases intestinal and portal blood flow, inhibits gastric acid secretion, and decreases intestinal motility, leading up to 20% decrease in PN provisions with treatment in patients with SBS. However, these agents can take weeks to months to take effect and is associated with known risk of developing intestinal growths and cancer that require ongoing surveillance with screening endoscopy. There is a need for other medications to help in the treatment of SBS.

Crofelemer is a novel anti-diarrheal drug that reduces intestinal chloride ion and fluid secretion. It is an FDA approved treatment for HIV-diarrhea (MytesiTM). Its anti-diarrheal properties are due to modulation of chloride ion channel secretion by cystic fibrosis transmembrane conductance regulator (CFTR) and/or Ca2+ activated Cl- channel (CaCC).

Crofelemer has been shown to be a dose-dependent, partial antagonism of CFTR and complete inhibition of CaCC without any changes in the intracellular cyclic Adenosin Monophosphate (cAMP) or calcium levels. Crofelemer also does not have any effects on gut motility or peristalsis. It also has been shown to have minimal absorptive capacity, therefore will not interact with other medications and limit serious adverse events.

It is unknown if Crofelemer can be effective in reducing diarrhea in patients with SBS. There have been case reports that suggest beneficial effects on nutritional status and improvement of diarrhea with tablets of Crofelemer in SBS. This study aims to assess the efficacy of Crofelemer in patients with SBS and ileostomy on Parenteral support.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must understand and provide written informed consent before they can participate in the study. They must understand the study procedures of the trial and be willing to complete the required assessments;
2. Male and female patients aged ≥ 18 years;
3. SBS patients without colon in continuity:
4. Patients with history of SBS resulting in intestinal failure caused by a major intestinal resection (e.g., injury, cancer, Crohn's disease, vascular disease, volvulus, intussusceptions or other causes). Diagnosis of SBS will be defined as remaining small bowel excluding colon in continuity and considered stable with regard to parenteral support (PS) need. Intestinal failure will be defined according to the recommendations of the American Society of Parenteral and Enteral Nutrition (ASPEN), i.e. a reduction of gut function below the minimum necessary for the absorption of macronutrients and/or water and electrolytes, such that intravenous (IV) supplementation is required to maintain health and/or growth;
5. At least 6 months elapsed since last surgical bowel resection;
6. No restorative surgery planned in the overall study period;
7. Patients with at least 6 continuous months of PS dependency (parenteral nutrition and/or intravenous fluids) before entry in the study;
8. Patients receiving stable PS (fluids, electrolytes or nutrients) at least three times per week to meet caloric, fluid or electrolytes needs with no major changes in provisions for at least 12 weeks;
9. Patients with Crohn's disease will have to be in clinical remission for ≥ 12 weeks before entry in the study;
10. Patients must be able to ingest solid or semi-solid foods and drink fluids;
11. If female and of child-bearing potential, the patient use a highly effective method of birth control for the entire study duration. Highly effective birth control methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence;
12. If female and of child-bearing potential, the patient must have a negative urine pregnancy test prior the first administration of the study drugs;
13. Male patients must agree to use an acceptable form of birth control during the study and for 30 days after the last dose;
14. Satisfactory general health status as determined by the investigator based on medical history and physical examination

Exclusion Criteria:

1. Body mass index (BMI) <17.5 or >30 kg/m2;
2. Presence of clinically significant intestinal adhesions and/or chronic abdominal pain that can interfere with the conduct of the study;
3. Presence of confirmed active infection, temperatures >100°Farenheit, or symptoms of an upper respiratory infection
4. Patients with Radiological (Radiography and/or CT) signs of significant bowel dilatation or pseudo-obstruction;
5. Active Crohn's disease as evaluated by standard procedures employed by the investigator;
6. Inflammatory bowel disease (IBD) that required immunosuppressant therapy that has been introduced or changed within last 3 months or treatment with biologics within the last 6 months;
7. Intestinal or other major surgery scheduled within the time frame of the study;
8. Visible blood in the stool within the last 3 months;
9. Ongoing radiation enteritis or the presence of damaged enteral tissue due to radiation enteritis, scleroderma, celiac disease, refractory or tropical sprue;
10. Compromised immune system (e.g., acquired immune deficiency syndrome [AIDS], severe combined immunodeficiency);
11. Inadequate hepatic function: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 upper limit of normal (ULN), total bilirubin >1.25 ULN or alkaline phosphatases >2.5 ULN;
12. Inadequate renal function: serum creatinine or blood urea nitrogen >1.5 ULN;
13. Urine sodium <20 mmol/day;
14. More than four SBS-related hospital admissions (unless one or more admissions were to rule out line sepsis) within the past 12 months or hospital admission within 1 month before screening;
15. Previous use of Crofelemer or potential allergies to Crofelemer or its constituents;
16. Use of infliximab, growth hormone or growth factors such as native glucagon-like peptide-2 (GLP-2) or other biological therapy within the last 12 weeks;
17. Current or past use of teduglutide within the last 3 months;
18. Use of systemic corticosteroids, methotrexate, cyclosporine, tacrolimus, sirolimus, octreotide, intravenous glutamine within the last 30 days;
19. If taken at screening, use of antimotility and antidiarrheal agents (loperamide, difenoxylate, codeine and other opiates), H2-receptor antagonists, proton pump inhibitors, bile sequestering agents, oral glutamine, diuretics and oral rehydration solutions is required to be at stable average weekly doses for at least 4 weeks prior to screening evaluations and to remain stable for the entire study duration;
20. Use of antibiotics within the last 30 days unless they were administered while ruling out line sepsis or for a dental procedure;
21. Alcohol or drug abuse within the last year;
22. Pregnant or lactating women;
23. History of any malignancy in the past 1 year;
24. History of psychiatric illnesses;
25. History of any other uncontrolled chronic or acute concomitant disease which, in the Investigator's opinion, would contraindicate study participation or confound interpretation of the results;
26. Patient not capable of understanding or not willing to adhere to the study visit schedules and other protocol requirements;
27. Participation in any other interventional clinical study within 30 days prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Ostomy output reduction | 12 weeks
  Change in ostomy output from baseline over the entire 12-week treatment period as average weekly ostomy output at week 12.

SECONDARY OUTCOMES:
Change in average weekly Parenteral Support (PS) volume | 16 weeks from treatment start
Change in SBS-QoL (Short bowel syndrome quality of life) | 16 weeks from treatment start
  Patient reported questionnaire with
Change in GSRS (Gastrointestinal Symptom Rating Scale) | 16 weeks from treatment start
Change in intestinal absorption of fluids and macronutrients with consequent reduction of macronutrient requirements in patients with SBS | 12 weeks after start or End of Trial
Change in weekly need for parenteral electrolytes | 16 weeks from treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Russell, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Plan to share unidentified data to Napo Pharmaceuticals Inc for future study planning